CLINICAL TRIAL: NCT00611325
Title: Phase II Trial of Avastin Plus Bortezomib for Patients With Recurrent Malignant Glioma
Brief Title: Phase II Avastin + Bortezomib for Patients With Recurrent Malignant Glioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00003596
Record Dates: First submitted 2008-01-28; First posted 2008-02-08 (Estimated); Results first posted 2014-02-04 (Estimated); Last update posted 2014-03-12 (Estimated); Status verified 2014-02

CONDITIONS: Glioblastoma; Gliosarcoma
Keywords: Glioblastoma; Gliosarcoma; Glioblastoma multiforme; Recurrent malignant glioma; GBM; Recurrent GBM; Malignant glioma; Brain tumor; Avastin; Bevacizumab; Bortezomib; Velcade
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Glioma; Brain Neoplasms | interventions — Bevacizumab; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EIAED (Experimental): Patients taking enzyme-inducing anti-epileptic drugs (EIAEDs). Avastin was administered intravenously at a dose of 15 mg/kg every 3 weeks. Bortezomib was adminstered intravenously at a dose of 2.5 mg/m2 on days 1, 4, 8, 11, 22, 25, 29, and 32 of a 42-day cycle.
  Interventions: Drug: Avastin; Drug: Bortezomib
- Non-EIAED (Experimental): Patients not taking enzyme-inducing anti-epileptic drugs (EIAEDs). Avastin was administered intravenously at a dose of 15 mg/kg every 3 weeks. Bortezomib was adminstered intravenously at a dose of 1.7 mg/m2 on days 1, 4, 8, 11, 22, 25, 29, and 32 of a 42-day cycle.
  Interventions: Drug: Avastin; Drug: Bortezomib

INTERVENTIONS:
Drug: Avastin — Avastin was administered intravenously at the dose 15 mg/kg every 3 weeks.
  Other Names: Bevacizumab
Drug: Bortezomib — Bortezomib was administered on days 1, 4, 8, 11, 22, 25, 29, & 32 of a 42-day cycle. Bortezomib was 1.7 mg/m2 for patients not taking EIAEDs & 2.5 mg/m2 for patients taking EIAEDs.
  Other Names: Velcade

SUMMARY:
Primary Objective To estimate 6-month progression free survival probability of patients with recurrent glioblastoma multiforme treated with bortezomib plus Avastin. This efficacy assessment will be made separately among patients on enzyme-inducing anti-epileptic drugs and non enzyme-inducing anti-epileptic drugs.

Secondary Objectives To evaluate safety & tolerability of bortezomib plus Avastin among patients with recurrent malignant glioma.

To evaluate radiographic response, progression free survival & overall survival of patients with recurrent malignant glioma treated with bortezomib plus Avastin

DETAILED DESCRIPTION:
This is an open-label, 2-arm Phase II study assessing safety & efficacy of bortezomib in combination with Avastin for patients with recurrent glioblastoma multiforme (gbm). 56 total patients with recurrent WHO grade IV malignant gliomas have been enrolled on study. Avastin was administered intravenously at a dose of 15 mg/kg every 3 weeks. Bortezomib was administered on days 1, 4, 8, 11, 22, 25, 29, & 32 of a 42-day cycle. The dose of bortezomib was 1.7 mg/m2 for non-EIAED patients & 2.5 mg/m2 for EIAED patients. Treatment continued until either evidence of progressive disease, unacceptable toxicity, non-compliance with study follow-up / withdrawal of consent. Brain MRIs were obtained after every cycle.

Bortezomib administration is associated with mild toxicity in most patients, such as fatigue, diarrhea & nausea, constipation & peripheral neuropathy. Less common, bortezomib administration leads to more significant hematologic toxicities & peripheral neuropathies. Most significant toxicities associated with Avastin in recently completed phase II clinical trial at Duke were thrombotic complications & grade 2 proteinuria. "Unacceptable" toxicities rates of 15 percent or less were considered desirable, while rates of 40 percent or greater were considered undesirable. The statistical hypothesis that needed testing differentiated between 15% & 40% rate of unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

Patients have histologically confirmed diagnosis of recurrent/progressive WHO grade IV malignant glioma (MG)

* Age >18 yrs
* No prior treatment with bortezomib, & no Avastin in last 3 months, not allowed to have progressed to Avastin regimen. No history of > or equal to grade 2 CNS hemorrhage or grade 3 or higher toxicities while on Avastin
* At least 6 weeks from surgical resection, 4 weeks from end of radiotherapy & enrollment in this study
* Karnofsky Performance Status (KPS) > or equal to 70%
* Hemoglobin (Hgb) > or = to 9 g/deciliter (dL), absolute neutrophil count (ANC) > or = to 1,500 cells/microliter, platelets > or = to 125,000 cells/microliter;
* Serum creatinine <1.5 mg/dL, serum glutamic oxalocetic transaminase (SGOT) & bilirubin <1.5 x upper limit of normal
* Signed informed consent approved by IRB;
* If sexually active, patients must agree to take contraceptive measures for duration of treatments
* May have had up to 3 biological therapies (such as tyrosine kinase inhibitors, topoisomerase I or II inhibitors, or rapamycin)

Exclusion Criteria:

* Gr 2 or greater peripheral neuropathy at time of study enrollment
* No prior taxanes, as it predisposes to sensory neuropathy
* Co-medication that may interfere with study results, e.g. immuno-suppressive agents other than corticosteroids
* Greater than 3 prior recurrences
* Evidence of CNS hemorrhage on baseline MRI on CT scan (except for grade 1 hemorrhage that has been stable for at least 3 months)
* History of thrombotic or hemorrhagic stroke or myocardial infarction within 6 months
* Requires therapeutic anti-coagulation
* At least 4 weeks from Day 0 of prior monthly chemotherapy (at least 6 weeks if a nitrosourea). At least 1 week from last dose of daily chemotherapy (such as metronomic temozolomide, cytoxan) or targeted therapies administered daily (such as gleevec, tarceva)
* Pregnancy or breast feeding
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection requiring IV antibiotics & psychiatric illness/social situations that would limit compliance with study requirements, or disorders associated with significant immunocompromised state
* Patients with another primary malignancy that has required treatment within past year.

Avastin-Specific Concerns:

* Any prior history of hypertensive crisis or hypertensive encephalopathy
* Systolic blood pressure (BP) > 150 mmHg or diastolic BP > 100 mmHg
* Unstable angina
* New York Heart Association Gr II or > congestive heart failure
* History of myocardial infarction within 6 months
* History of stroke within 6 months
* Clinically significant peripheral vascular disease
* Evidence of bleeding diathesis, coagulopathy as documented by an elevated prothrombin time (PT), partial thromboplastin time (PTT)/bleeding time
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 0, anticipation of need for major surgical procedure during course of study
* Minor surgical procedures, fine needle aspirations or core biopsies within 7 days prior to Day 0
* Urine protein: creatinine ratio > or = to 1.0 at screening
* History of abdominal fistula, GI perforation, or intra-abdominal abscess within 6 months prior to Day 0
* Serious, non-healing wound, ulcer, or bone fracture
* Known hypersensitivity to any component of Avastin
* Inability to comply with study and/or follow-up procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2008-05; Primary Completion 2009-09 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine B Peters, MD, Principal Investigator — Duke Health
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

REFERENCES:
- See also: The Preston Robert Tisch Brain Tumor Center at DUKE — http://www.cancer.duke.edu/btc/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | EIAED | Non-EIAED
Started | 28 | 28
Completed | 28 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EIAED | Non-EIAED | Total
Number analyzed (Participants) | 28 | 28 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.73 (12.57) | 55.03 (11.36) | 53.88 (11.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 12 | 20
  Male | 20 | 16 | 36
Region of Enrollment [Number; unit: participants]
  United States | 28 | 28 | 56

OUTCOME MEASURES:

1. Primary Outcome: 6-month Progression-free Survival (PFS)
Description: Percentage of participants surviving six months from the initiation of treatment without progression of disease. PFS was defined as the time from the initiation of treatment to the date of the first documented progression according to the Macdonald criteria, or to death due to any cause. Per Macdonald, progression is a ≥ 25% increase in the sum of the products of perpendicular diameters of enhancing lesions, any new lesion or clinical deterioration.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | EIAED | Non-EIAED
Number analyzed (Participants) | 28 | 28
percentage of participants | 25 [9.0 to 41.0] | 28.6 [11.9 to 45.3]

2. Secondary Outcome: Median Progression Free Survival (PFS)
Description: Time in months from the start of study treatment to the date of first progression according to Macdonald criteria, or to death due to any cause. Per Macdonald, progression is a ≥ 25% increase in the sum of the products of perpendicular diameters of enhancing lesions, any new lesion, or clinical deterioration. Patients alive who had not progressed as of the last follow-up had PFS censored at the last follow-up date. Median PFS was estimated using a Kaplan-Meier curve.
Time Frame: Time in months from the start of study treatment to the date of first progression or death. Assessed up to 60 months.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | EIAED | Non-EIAED
Number analyzed (Participants) | 28 | 28
months | 2 [2 to 4] | 2.5 [1 to 4]

3. Secondary Outcome: Median Overall Survival (OS)
Description: Time in months from the start of study treatment to the date of death. Patients alive as of the last follow-up had OS censored at the last follow-up date. Median OS was estimated using a Kaplan-Meier curve.
Time Frame: Time in months from the start of study treatment to date of death due to any cause. Assessed up to 60 months.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | EIAED | Non-EIAED
Number analyzed (Participants) | 28 | 28
months | 8 [5 to 11] | 6 [4 to 10]

4. Secondary Outcome: Radiographic Response Rate
Description: The percentage of participants with a complete or partial response at any assessment as determined by the Macdonald criteria. A confirmation of response was not required. Per Macdonald criteria, complete response (CR) was the disappearance of all target lesions and partial response (PR) was a ≥50% decrease in the sum of the longest diameter of target lesions, no new lesions and stable or decreasing steroid dose. Objective response =CR+PR. Tumor assessments were done at baseline and at the end of each 6 week treatment cycle, and overall best response was recorded.
Time Frame: 60 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | EIAED | Non-EIAED
Number analyzed (Participants) | 28 | 28
percentage of participants | 7.1 [0 to 16.6] | 39.3 [21.2 to 57.4]

5. Secondary Outcome: Number of Patients With Grade 3 or Greater, Treatment-related, Non-hematologic Toxicities
Description: Number of patients with grade 3 or greater, treatment-related, non-hematologic toxicities based on Common Terminology Criteria for Adverse Events (CTCAE) version 3.0.
Time Frame: 60 months
Measure: Number; unit: participants
Arm/Group | EIAED | Non-EIAED
Number analyzed (Participants) | 28 | 28
participants | 27 | 24

ADVERSE EVENTS:
Time Frame: 60 months
Description: The adverse events for this study were collected using Common Terminology Criteria for Adverse Events (CTCAE) version 3.0, and have been converted to CTCAE version 4.0 for entry into ClinicalTrials.gov.
Groups:
- EIAED: Avastin: Avastin was administered intravenously at the dose 15 mg/kg every 3 weeks.
  Bortezomib: Bortezomib was administered on days 1, 4, 8, 11, 22, 25, 29, & 32 of a 42-day cycle. Bortezomib was 2.5 mg/m2 for patients taking EIAEDs.
- Non-EIAED: Avastin: Avastin was administered intravenously at the dose 15 mg/kg every 3 weeks.
  Bortezomib: Bortezomib was administered on days 1, 4, 8, 11, 22, 25, 29, & 32 of a 42-day cycle. Bortezomib was 1.7 mg/m2 for patients not taking EIAEDs.
Arm/Group | EIAED | Non-EIAED
Serious Adverse Events (participants affected / at risk) | 11/28 | 5/28
Other Adverse Events (participants affected / at risk) | 28/28 | 28/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EIAED (N=28) | Non-EIAED (N=28)
Anemia (Blood and lymphatic system disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 2 | 1
Fatigue (General disorders) | 1 | 0
Fever (General disorders) | 2 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 2
Fracture (Injury, poisoning and procedural complications) | 2 | 0
Platelet count decreased (Investigations) | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 2
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Ataxia (Nervous system disorders) | 3 | 2
Cognitive disturbance (Nervous system disorders) | 1 | 1
Hydrocephalus (Nervous system disorders) | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 2 | 0
Syncope (Nervous system disorders) | 0 | 1
Confusion (Psychiatric disorders) | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 1
Thromboembolic event (Vascular disorders) | 2 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EIAED (N=28) | Non-EIAED (N=28)
Anemia (Blood and lymphatic system disorders) | 2 | 2
Blurred vision (Eye disorders) | 1 | 3
Extraocular muscle paresis (Eye disorders) | 2 | 0
Eye disorders - Other, specify (Eye disorders) | 0 | 3
Eye pain (Eye disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 13 | 6
Constipation (Gastrointestinal disorders) | 3 | 8
Diarrhea (Gastrointestinal disorders) | 13 | 11
Fecal incontinence (Gastrointestinal disorders) | 1 | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 3 | 4
Hemorrhoids (Gastrointestinal disorders) | 0 | 1
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 5 | 6
Nausea (Gastrointestinal disorders) | 12 | 7
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Stomach pain (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 9 | 5
Edema limbs (General disorders) | 2 | 6
Fatigue (General disorders) | 18 | 21
Fever (General disorders) | 2 | 2
Gait disturbance (General disorders) | 3 | 5
Non-cardiac chest pain (General disorders) | 0 | 1
Pain (General disorders) | 1 | 2
Device related infection (Infections and infestations) | 1 | 0
Eye infection (Infections and infestations) | 0 | 1
Infections and infestations - Other, specify (Infections and infestations) | 2 | 6
Kidney infection (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 2
Skin infection (Infections and infestations) | 1 | 0
Tooth infection (Infections and infestations) | 0 | 1
Upper respiratory infection (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 2 | 5
Alanine aminotransferase increased (Investigations) | 0 | 3
Alkaline phosphatase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 1
Lipase increased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 5 | 6
Platelet count decreased (Investigations) | 11 | 14
Weight loss (Investigations) | 1 | 1
White blood cell decreased (Investigations) | 3 | 8
Anorexia (Metabolism and nutrition disorders) | 1 | 10
Dehydration (Metabolism and nutrition disorders) | 4 | 5
Hyperglycemia (Metabolism and nutrition disorders) | 4 | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 3 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 10 | 13
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 | 4
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 | 3
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 4
Ataxia (Nervous system disorders) | 13 | 9
Cognitive disturbance (Nervous system disorders) | 4 | 6
Depressed level of consciousness (Nervous system disorders) | 4 | 7
Dizziness (Nervous system disorders) | 3 | 2
Dysphasia (Nervous system disorders) | 4 | 4
Headache (Nervous system disorders) | 7 | 9
Memory impairment (Nervous system disorders) | 1 | 5
Nervous system disorders - Other, specify (Nervous system disorders) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 4
Peripheral sensory neuropathy (Nervous system disorders) | 18 | 15
Seizure (Nervous system disorders) | 7 | 11
Syncope (Nervous system disorders) | 0 | 2
Tremor (Nervous system disorders) | 1 | 2
Trigeminal nerve disorder (Nervous system disorders) | 0 | 1
Agitation (Psychiatric disorders) | 1 | 3
Anxiety (Psychiatric disorders) | 0 | 4
Confusion (Psychiatric disorders) | 4 | 5
Depression (Psychiatric disorders) | 2 | 5
Insomnia (Psychiatric disorders) | 1 | 5
Personality change (Psychiatric disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 3 | 4
Urinary incontinence (Renal and urinary disorders) | 1 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 6
Hypertension (Vascular disorders) | 5 | 6
Hypotension (Vascular disorders) | 3 | 2
Thromboembolic event (Vascular disorders) | 4 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No